CLINICAL TRIAL: NCT03458364
Title: Comparison of High Flow Nasal Cannula With Noninvasive Ventilation in Facilitating Weaning Chronic Obstructive Pulmonary Disease From Invasive Ventilation: a Prospective Randomized Controlled Study
Brief Title: Comparison of HFNC With NIV in Weaning COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jie Li (Other)
Collaborators: Binzhou Medical University (Other)
Responsible Party: Sponsor-Investigator, Jie Li, Clinical education coordinator, Rush University Medical Center
Organization: Rush University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HFNC-002
Record Dates: First submitted 2018-03-02; First posted 2018-03-08 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Chronic Obstructive Pulmonary Disease With (Acute) Exacerbation
Keywords: Weaning; Noninvasive ventilation; High flow nasal cannula
MeSH Terms: interventions — Noninvasive Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High flow nasal cannula (Experimental): High flow nasal cannula (HFNC) is a type of oxygen device, which provides high concentration oxygen in a high flow, which exceeds patient's inspiratory flow demand, to improve oxygenation.
  Interventions: Device: High flow nasal cannula
- Noninvasive ventilation (Active Comparator): Non-invasive ventilation (NIV) refers to the provision of ventilatory support through the patient's upper airway using a mask. This technique is distinguished from those which bypass the upper airway with a tracheal tube, laryngeal mask, or tracheostomy and are therefore considered invasive.
  Interventions: Device: Noninvasive ventilation

INTERVENTIONS:
Device: High flow nasal cannula — High-flow nasal cannula (HFNC) oxygen therapy is a recent technique delivering a high flow of heated and humidified gas. HFNC is simpler to use and apply than noninvasive ventilation (NIV) and appears to be a good alternative treatment for hypoxemic acute respiratory failure (ARF). HFNC is better tolerated than NIV, delivers high fraction of inspired oxygen (FiO2), generates a low level of positive pressure and provides washout of dead space in the upper airways, thereby improving mechanical pulmonary properties and unloading inspiratory muscles during ARF.
  Other Names: High flow high humidity nasal cannula
  Arms: High flow nasal cannula
Device: Noninvasive ventilation — Non-invasive ventilation (NIV) is the use of airway support administered through a face (nasal) mask instead of an endotracheal tube. Inhaled gases are given with positive end-expiratory pressure often with pressure support or with assist control ventilation at a set tidal volume and rate. Numerous studies have shown this technique to be as effective as, and better tolerated than, intubation and mechanical ventilation in patients with exacerbations of COPD
  Other Names: Noninvasive positive pressure ventilation; Noninvasive mechanical ventilation
  Arms: Noninvasive ventilation

SUMMARY:
High flow nasal cannula (HFNC) has been shown to improve oxygenation and facilitate weaning in hypoxemia patients. Some clinical studies show the benefits of using HFNC in COPD patients, including reducing dead space and work of breathing. However, no clinical study has been to investigate the value of HFNC in weaning COPD patients from invasive ventilation. Thus, we proposed a randomized controlled trial to compare the use of HFNC and noninvasive ventilation (NIV) in weaning COPD.

DETAILED DESCRIPTION:
High flow nasal cannula (HFNC) provides high concentration oxygen in a high flow, which exceeds patient's inspiratory flow demand, to improve oxygenation. In a recent meta-analysis of seven trials with 1771 patients, HFNC was shown to improve oxygenation and avoid intubation in patients with severe hypoxemia. The high velocity of the gas can rinse the dead space of the upper airway and reduce CO2 rebreathing, reduce COPD patients' work of breathing and improve the dynamic compliance of respiratory system.

Thus, we proposed a randomized controlled trial to investigate the value of high flow nasal cannula in weaning AECOPD patients from invasive ventilation, with comparison of noninvasive ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Intubated patients with Chronic obstructive pulmonary disease exacerbation
* Meeting extubation criteria (Pulmonary infection control window)
* Age > 21years and < 90 years

Exclusion Criteria:

* Tracheotomy
* Combined with severe dysfunction of other organs, including heart, brain, liver, and renal failure;
* Hemodynamic instability
* Contraindication to NIV: cannot use mask, such as facial injury, burns or deformities; cannot cooperate with NIV such as delirium; copious secretions with weak cough ability; gastric over distention, and vomiting;
* Contraindication to HFNC: rhinitis, nasal congestion, deformities or blockage.
* Weak cough ability with copious secretions
* Refuse to participate in the study

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
pH | change from the baseline pH within 48 hours
  pH
PaCO2 | change from the baseline PaCO2 within 48 hours
  PaCO2 in mmHg
PaO2/FiO2 | change from the baseline PaO2/FiO2 within 48 hours
  partial pressure of oxygen in arterial blood/ fraction of inspired oxygen in mmHg
HR | change from the baseline HR within 48 hours
  Heart Rate in beats per minute
MAP | change from the baseline MAP within 48 hours
  mean arterial pressure in mmHg
RR | change from the baseline RR within 48 hours
  respiratory rate in breaths per minute

SECONDARY OUTCOMES:
duration of respiratory support | 28 days
  hours of ventilator use
Length of ICU stay | 28 days
  Days of stay in ICU
Mortality | 28 days
the patients' comfort score | 48 hours
  comfort score of using high flow nasal cannula or noninvasive ventilator, ranging from 1 to 10. 1 means very comfortable, 10 means very uncomfortable.
incidence of nasal trauma | 28 days
incidence of barotrauma | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Xiaozhi Wang, MD, Study Chair — Binzhou Medical University
Locations (1):
- Binzhou Medical University Hospital, Yantai, Shandong, China

REFERENCES:
- [Background] Zhu Y, Yin H, Zhang R, Wei J. High-flow nasal cannula oxygen therapy versus conventional oxygen therapy in patients with acute respiratory failure: a systematic review and meta-analysis of randomized controlled trials. BMC Pulm Med. 2017 Dec 13;17(1):201. doi: 10.1186/s12890-017-0525-0. PMID 29237436
- [Background] Mauri T, Turrini C, Eronia N, Grasselli G, Volta CA, Bellani G, Pesenti A. Physiologic Effects of High-Flow Nasal Cannula in Acute Hypoxemic Respiratory Failure. Am J Respir Crit Care Med. 2017 May 1;195(9):1207-1215. doi: 10.1164/rccm.201605-0916OC. PMID 27997805
- [Background] Lv Y, Lv Q, Lv Q, Lai T. Pulmonary infection control window as a switching point for sequential ventilation in the treatment of COPD patients: a meta-analysis. Int J Chron Obstruct Pulmon Dis. 2017 Apr 24;12:1255-1267. doi: 10.2147/COPD.S126736. eCollection 2017. PMID 28490869
- [Background] Rochwerg B, Brochard L, Elliott MW, Hess D, Hill NS, Nava S, Navalesi P Members Of The Steering Committee, Antonelli M, Brozek J, Conti G, Ferrer M, Guntupalli K, Jaber S, Keenan S, Mancebo J, Mehta S, Raoof S Members Of The Task Force. Official ERS/ATS clinical practice guidelines: noninvasive ventilation for acute respiratory failure. Eur Respir J. 2017 Aug 31;50(2):1602426. doi: 10.1183/13993003.02426-2016. Print 2017 Aug. PMID 28860265